CLINICAL TRIAL: NCT00005586
Title: A UKCCCR Study of Adjuvant Chemotherapy for Colorectal Cancer
Brief Title: Leucovorin and Fluorouracil Compared With Observation in Treating Patients With Colorectal Cancer That Has Been Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067660; NCRI-QUASAR1; EU-99053; UKCCCR-QUASAR1; ISRCTN82375386
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-03

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Leucovorin; Fluorouracil; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: L-leucovorin
Drug: fluorouracil
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether chemotherapy is more effective than observation in patients who have had surgery to remove colorectal cancer.

PURPOSE: This randomized phase III trial is studying leucovorin and fluorouracil to see how well they work compared to observation in treating patients with colorectal cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare all-cause mortality in patients with resected colorectal cancer treated with adjuvant chemotherapy with L-leucovorin and fluorouracil vs observation.
* Compare the recurrence rates in patients treated with this regimen vs observation.
* Compare the effectiveness of a monthly 5-day schedule vs a once weekly schedule of L-leucovorin and fluorouracil in this patient population.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to receive adjuvant chemotherapy (arm I) or undergo observation only (arm II).

* Arm I: Within 12 weeks of surgery, patients receive L-leucovorin IV followed by fluorouracil IV on days 1-5 every 4 weeks for 6 courses. Alternatively, patients may receive L-leucovorin IV followed by fluorouracil IV on day 1 weekly for 30 weeks.
* Arm II: Patients undergo observation. Patients are followed annually.

PROJECTED ACCRUAL: A total of 2,500 patients (1,250 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Completely resected stage II or III colorectal cancer
* No distant metastases
* No positive resection margins
* No positive peritoneal washings

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No clear definite indication for, or contraindication against, systemic chemotherapy with L-leucovorin and fluorouracil

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy in observation only arm

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent radiotherapy allowed in adjuvant chemotherapy arm provided chemotherapy administered on the once weekly schedule

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 1997-10

PRIMARY OUTCOMES:
All-cause mortality

SECONDARY OUTCOMES:
Death from colorectal cancer
Disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Norman Williams, MD, Study Chair — Royal London Hospital
Locations (1):
- Royal London Hospital, London, England, United Kingdom

REFERENCES:
- [Result] Quasar Collaborative Group; Gray R, Barnwell J, McConkey C, Hills RK, Williams NS, Kerr DJ. Adjuvant chemotherapy versus observation in patients with colorectal cancer: a randomised study. Lancet. 2007 Dec 15;370(9604):2020-9. doi: 10.1016/S0140-6736(07)61866-2. PMID 18083404